CLINICAL TRIAL: NCT04152668
Title: Non-surgical Treatment of Peri-implantitis With and Without Erythritol Air-polishing: A 12-month Randomized Controlled Trial
Brief Title: Non-surgical Treatment of Peri-implantitis With and Without Erythritol Air-polishing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Knut N. Leknes (Other)
Responsible Party: Sponsor-Investigator, Knut N. Leknes, Professor, University of Bergen
Organization: University of Bergen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UiB, IKO 2019
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis; Air-polishing; Erythritol
MeSH Terms: conditions — Peri-Implantitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Randomized, single-masked controlled trial (RCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Forty patients diagnosed with peri-implantitis on at least one implant will be randomly allocated by tossing a coin into test or control group. Two different operators will participate in the study (ML and AS). ML masked to the treatment assignment, will collect the data, and AS will perform the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium curette and ultrasonic. (Active Comparator): Control implants will be debrided with titanium curette and ultrasonic device without time limit.
  Interventions: Procedure: Titanium curette.; Procedure: Ultrasonic
- Titanium curette, ultrasonic and air-polishing. (Experimental): Test implants will be treated with titanium curette, ultrasonic device and a specially designed nozzle mounted on a hand piece (Perio-Flow) connected to an airflow unit also without time limit.
  Interventions: Procedure: Titanium curette.; Procedure: Ultrasonic; Procedure: Air-polishing

INTERVENTIONS:
Procedure: Titanium curette. — Implant debridement.
Procedure: Ultrasonic — Implant debridement.
  Other Names: Ultrasonic device
Procedure: Air-polishing — Implant debridement and polishing.
  Other Names: Air-polishing device
  Arms: Titanium curette, ultrasonic and air-polishing.

SUMMARY:
Erythritol is a natural sugar alcohol (a four-carbon polyol) produced by the reduction of erythrose. It is considered safe as food additive and has many of the functional properties that are important for subgingival debridement. Current evidence includes no prospective studies comparing the outcomes of a low abrasive erythritol air-polishing as an adjunctive therapy to conventional titanium and ultrasonic debridement of patients in a maintenance program with peri-implantitis. Thus, the main purpose of this randomized, single-masked controlled trial (RCT) is to assess whether low abrasive erythritol air-polishing has an adjunct effect to conventional non-surgical treatment of peri-implantitis.

DETAILED DESCRIPTION:
This RCT will enroll subjects among patients in need for non-surgical treatment of peri-implantitis at a private dental clinic in Stavanger, Norway. Forty patients diagnosed with peri-implantitis on at least one implant will be randomly allocated by tossing a coin into test or control group. Patients with cement-retained and screw-retained supraconstructions will be included.

Treatment of peri-implantitis will be performed by one operator (AS) at baseline, 3-, 6-, 9- and 12-month follow-up visits. Local anesthesia will be used when needed. In the test group, implants will be treated with titanium curette, ultrasonic device and a specially designed nozzle mounted on a hand piece (Perio-Flow) connected to an airflow unit.

In the control group, implant with peri-implantitis will be debrided with titanium curette and ultrasonic device only. Test and control debridement will be performed without time limit. The treatment will continue until the operator is judging the implant surface to be free for supra- and subgingival deposits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 20 - 85 years who have received one or more dental implant(s) being in successful function for more than 12 months and restored with an optimal supraconstruction
* Diagnosed with peri-implantitis based on the following criteria:

  * Bleeding and/or suppuration upon gentle probing
  * Increased probing depths (PD) compared with previous examinations or PD of ≥ 4 mm in at least one site around the implant
  * Crestal bone level (CBL) loss ≥2 mm compared with baseline registration

Exclusion Criteria:

* Surgical treatment of peri-implantitis the last 6 months
* Supportive periodontal therapy within 3 months
* Use of systemic antibiotic within 6 months
* A history of non-compliant behavior
* Inflammation around implant without evidence of bone loss
* Periapical peri-implantitis
* Subjects with implant fracture, ceramic implants, or detectable subgingival cement
* Any current medical condition affecting the use of the abrasive air-polishing device.
* Subjects with diabetes mellitus, cancer, HIV/aids, acute infections, liver or kidney dysfunction/failure,
* Current pregnancy or breastfeeding

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in probing depth (PD) | 12 moths
  PD as the distance in mm from the implant mucosal margin to the probable base of the pocket at six sites;
Crestal bone level (CBL) | 12 months
  Intraoral digitalized radiographs will be taken with customized Eggen-holder and long cone, parallel technique to assess CBL. The distance from implant platform to the mesial and distal bone levels will be measured by using the software program DIGORA (Soredex, Helsinki).

SECONDARY OUTCOMES:
Bleeding on probing (BoP) | 12 months
  BoP as the presence of bleeding after gentle probing (Renvert et al. 2017).
Gingival crevicular fluid (GCF) | 12 months
  Sample sites will be isolated with cottons rolls, carefully cleaned for supragingival plaque and air-dried. A perio paper strip will then be gently placed one to two mm into the entrance of the pocket and left in place for 30 seconds.
Visual analogue scale (VAS) | 12 months
  The scorings will be performed following completion of the debridement at baseline and at 6 and 12 months with 0 = "no pain" and 100 = "worst pain I can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Knut N. Leknes, Professor, Principal Investigator — Department of Clinical Dentistry - Periodontics, University of Bergen, NORWAY
Locations (1):
- Knut N. Leknes, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citations to publications related to the protocol: Background and Material and Methods.
- [Derived] Selimovic A, Bunaes DF, Lie SA, Lobekk MA, Leknes KN. Non-surgical treatment of peri-implantitis with and without erythritol air-polishing a 12-month randomized controlled trial. BMC Oral Health. 2023 Apr 24;23(1):240. doi: 10.1186/s12903-023-02973-5. PMID 37095488